CLINICAL TRIAL: NCT01404039
Title: Investigating Motor Cortex Processing for Pain Modulation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was halted due to lack of funding.
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010-p-001256
Record Dates: First submitted 2011-06-29; First posted 2011-07-27 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Motor Activity
Keywords: learning; pain perception
MeSH Terms: conditions — Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: There are 5 experiments: motor learning (3 groups, crossover), sensory learning (4 groups, parallel), observational task (2 groups, parallel), mental imagery (2 groups, parallel), and tDCS over the motor cortex (2 groups, crossover). Please note that the tDCS experiment has never been conducted.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (13):
- Motor Learning (ML) sighted (Experimental): In this arm, subject will perform motor Learning with visual feedback - ML sighted.
  There will be an anticipated total of 15 subjects in this experimental arm. This arm will be conducted as a cross-over design. The subjects will undergo the three interventions listed (motor learning with visual feedback, motor learning without visual feedback, and control group) in a counterbalanced randomized order. There will be at least 24 hours between each experimental session.
  Interventions: Behavioral: Motor Learning
- Motor Learning (ML) blind (Experimental): In this arm, subject will perform motor Learning without visual feedback - ML blind.
  There will be an anticipated total of 15 subjects in this experimental arm. This arm will be conducted as a cross-over design. The subjects will undergo the three interventions listed (motor learning with visual feedback, motor learning without visual feedback, and control group) in a counterbalanced randomized order. There will be at least 24 hours between each experimental session.
  Interventions: Behavioral: Motor Learning
- Motor Learning (ML) control group (Placebo Comparator): In this arm, subject will perform simple hand movements - control group. There will be an anticipated total of 15 subjects in this experimental arm. This arm will be conducted as a cross-over design. The subjects will undergo the three interventions listed (motor learning with visual feedback, motor learning without visual feedback, and control group) in a counterbalanced randomized order. There will be at least 24 hours between each experimental session.
  Interventions: Behavioral: Motor Learning
- Somatosensory Learning (SL sighted) (Experimental): In this arm, subject will perform sensory Learning with visual feedback - SL sighted.
  There will be an anticipated total of 10 subjects in this experimental arm. This experimental arm will be conducted in a parallel design with 4 groups (SL sighted, SL blind, Sactivation, SL control).
  Interventions: Behavioral: Somatosensory Learning
- Somatosensory Learning (SL blind) (Experimental): In this arm, subject will perform sensory Learning without visual feedback - SL blind.
  There will be an anticipated total of 10 subjects in this experimental arm. This experimental arm will be conducted in a parallel design with 4 groups (SL sighted, SL blind, Sactivation, SL control).
  Interventions: Behavioral: Somatosensory Learning
- Somatosensory Activation (S activation) (Experimental): In this arm, subject will receive simple sensory stimulation over their left index finger - Sactivation.
  There will be an anticipated total of 10 subjects in this experimental arm.This experimental arm will be conducted in a parallel design with 4 groups (SL sighted, SL blind, Sactivation, SL control).
  Interventions: Behavioral: Somatosensory Learning
- Somatosensory Learning (SL) control group (Placebo Comparator): In this arm,the subjects will not receive any somatosensory input (SL control group).
  There will be an anticipated total of 10 subjects in this experimental arm. This experimental arm will be conducted in a parallel design with 4 groups (SL sighted, SL blind, Sactivation, SL control).
  Interventions: Behavioral: Somatosensory Learning
- Observational Task (OT) - real (Experimental): In this arm, the subjects will perform an observational task - observation of hand movements. This experimental arm will be conducted in a parallel design. There will be 15 subjects per intervention.
  Interventions: Behavioral: Observational Task
- Observational Task (OT) - control group (Placebo Comparator): In this arm, the subjects will perform a controlled observational task - observation of geometric shapes. This experimental arm will be conducted in a parallel design. There will be 15 subjects per intervention.
  Interventions: Behavioral: Observational Task
- Mental Imagery (MI) - real (Experimental): In this arm, the subjects will perform mental imagery - mental imagery of finger movements. This experimental arm will be conducted in a parallel design. There will be 15 subjects per intervention.
  Interventions: Behavioral: Mental Imagery
- Mental Imagery (MI) - control group (Placebo Comparator): In this arm, the subjects will perform a controlled task - simple mental calculation. This experimental arm will be conducted in a parallel design. There will be 15 subjects per intervention.
  Interventions: Behavioral: Mental Imagery
- transcranial direct current stimulation - tDCS real (Experimental): tDCS will be applied over the motor cortex for 20minutes at an intensity of 2mA. 15 subjects will be enrolled. The subjects will undergo two interventions, real and sham in a counterbalanced randomized order. There will be at least 3 days between each experimental session.
  Interventions: Device: transcranial direct current stimulation
- transcranial direct current stimulation - tDCS sham (Placebo Comparator): tDCS will be applied over the motor cortex for 20minutes at an intensity of 2mA. The stimulation will be stopped after 30seconds.
  15 subjects will be enrolled. The subjects will undergo two interventions, real and sham in a counterbalanced randomized order. There will be at least 3 days between each experimental session.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Behavioral: Motor Learning — Subject will have to draw a set of shapes and words during 20 minutes.
  Arms: Motor Learning (ML) blind; Motor Learning (ML) control group; Motor Learning (ML) sighted
Behavioral: Somatosensory Learning — Subjects will perform a learning task involving sensory activation of the hand. The task will consist of learning letters of Braille.
  Arms: Somatosensory Activation (S activation); Somatosensory Learning (SL blind); Somatosensory Learning (SL sighted); Somatosensory Learning (SL) control group
Behavioral: Observational Task — Subjects will watch a 10 second video of a right-handed person performing movements of their left index finger. Subjects will be instructed to watch the video without any other specific instruction.
  Arms: Observational Task (OT) - control group; Observational Task (OT) - real
Behavioral: Mental Imagery — Subjects will be asked to perform mental imagery of motor practice - finger movements of the left hand for 10 minutes.
  Arms: Mental Imagery (MI) - control group; Mental Imagery (MI) - real
Device: transcranial direct current stimulation — Subjects will undergo active and sham tDCS stimulation in a randomized and counterbalanced order. During both active and sham stimulation, we will use electrodes of 35cm^2, intensity of 2mA for a duration of 20 minutes. The anode electrode will be placed over the right primary motor cortex (M1) and the cathode will be placed over the contralateral supraorbital area. For active stimulation, the current will be on for the duration of 20 minutes. For sham stimulation, the current will ramp up, and then down again for 30 seconds to simulate the sensation of active tDCS.
  Arms: transcranial direct current stimulation - tDCS real; transcranial direct current stimulation - tDCS sham

SUMMARY:
The purpose of this study is to investigate the effects of different types of interventions (motor learning, somatosensory learning, observation task, mental imagery and tDCS) on the perception of pain and motor cortex excitability in healthy male subjects. This is an exploratory study of healthy subjects only.

DETAILED DESCRIPTION:
There are 5 experiments:

Exp1: motor learning (3 groups, crossover) - motor leaning with and without visual feedback and a control group.

Exp2: sensory learning (4 groups, parallel) - sensory learning with and without feedback, an simple activation task and a control group.

Exp3: observational task (2 groups, parallel) - an motor observational task and a control group.

Exp4: mental imagery (2 groups, parallel) - a motor mental imagery and a control group.

Exp5: tDCS over the motor cortex (2 groups, crossover) - active and sham tDCS. Note that this study has never been completed.

ELIGIBILITY:
Inclusion Criteria

1. Provide informed consent to participate in the study
2. 18 to 64 years old
3. No presence of rheumatologic disease as self reported
4. No clinically significant or unstable medical or psychiatric disorder as self reported
5. No history of alcohol or substance abuse within the last 6 months as self reported
6. No neuropsychiatric co-morbidity as self reported
7. No Contraindications to single pulse TMS (TMS will be used to measure cortical excitability)

   * history of seizures
   * unexplained loss of consciousness
   * metal in the head
   * frequent or severe headaches or neck pain
   * implanted brain medical devices
8. No Contraindications to tDCS

   * metal in the head
   * implanted brain medical devices

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital (SRH)
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Motor Learning - MLsighted/MLblind/MLcontrol; Motor Learning (ML) MLblind/MLcontrol/MLsighted; Motor Learning (ML) MLcontrol Group/MLsighted/MLblind: This arm will be conducted as a cross-over design. The subjects will undergo the three interventions listed (motor learning with visual feedback, motor learning without visual feedback, and control group) in a counterbalanced randomized order. There will be at least 24 hours between each experimental session.
- Observational Task (OT): Observational Task: Subjects in this group will watch a 10 second video of a right-handed person performing movements of their left index finger at a 1 Hz rate on a screen at a distance of 1 meter away. Subjects will be instructed to watch the video without any other specific instruction.
- Observational Task (OT) - Control Group: Control Group -- Observational Task: Subjects in this group will be asked to watch a video of random geometric forms for the same duration of time as those in the observational task group.
- Mental Imagery (MI): Mental Imagery: Subjects will be seated in a chair and are asked to keep their arm and hand muscles fully relaxed. Then they will be asked to imagine repetitive movement of the left index finger to the left thumb for 5 minutes. Subjects then will be asked to imagine sequential movement of left finger to left thumb (thumb to 2nd, 3rd, 4th, 5th) for 5 minutes.
- Mental Imagery (MI) - Control Group: Control Group - Mental Imagery: Subjects will be asked to perform simple mental math calculations for 20 minutes. (ex. adding or subtracting a one digit number from a starting number (1+1=2; 2+1=3; 3+1= 4 and so on.)
- tDCS - Active; tDCS - Sham: This experimental arm will be conducted in a cross-over design (active tDCS and sham tDCS).
Period: Overall Study
Arm/Group | Motor Learning - MLsighted/MLblind/MLcontrol | Motor Learning (ML) MLblind/MLcontrol/MLsighted | Motor Learning (ML) MLcontrol Group/MLsighted/MLblind | Somatosensory Learning (SL Sighted) | Somatosensory Learning (SL Blind) | Somatosensory Activation (S Activation) | Somatosensory Learning (SL) Control Group | Observational Task (OT) | Observational Task (OT) - Control Group | Mental Imagery (MI) | Mental Imagery (MI) - Control Group | tDCS - Active | tDCS - Sham
Started | 5 | 5 | 5 | 10 | 10 | 10 | 10 | 15 | 15 | 15 | 15 | 0 | 0
Completed | 4 | 5 | 5 | 10 | 10 | 10 | 10 | 15 | 15 | 14 | 14 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Motor Learning (ML): This arm will be conducted as a cross-over design. The subjects will undergo the three interventions listed (motor learning with visual feedback, motor learning without visual feedback, and control group) in a counterbalanced randomized order. There will be at least 24 hours between each experimental session.
- Total: Total of all reporting groups
Arm/Group | Motor Learning (ML) | Somatosensory Learning (SL Sighted) | Somatosensory Learning (SL Blind) | Somatosensory Activation (S Activation) | Somatosensory Learning (SL) Control Group | Observational Task (OT) - Real | Observational Task (OT) - Control | Mental Imagery (MI) - Real | Mental Imagery (MI) - Control | Total
Number analyzed (Participants) | 15 | 10 | 10 | 10 | 10 | 15 | 15 | 15 | 15 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 10 | 10 | 10 | 10 | 15 | 15 | 15 | 15 | 115
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 10 | 10 | 10 | 10 | 15 | 15 | 15 | 15 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Cortex Excitability MEP Amplitude
Description: We aim to assess the effects of the intervention (ML, SL, OT and MI) on motor cortex excitability as measured by the change in motor evoked potential (using transcranial magnetic stimulation) before and after the given intervention.
  * For ML: MEP will be measured before and after each ML sessions in the same subject (crossover design - ML sighted/MLblind/ML control).
  * For SL: MEP will be measured before and after the treatment session in the each groups (parallel design - 1 session per group).
  * For OT: MEP will be measured before and after the treatment session in the each groups (parallel - 1 session per group).
  * For MI: MEP will be measured before and after the treatment session in the each groups (parallel design - 1 session per group).
Time Frame: after each intervention
Population: ML: crossover design - ML sighted/MLblind/ML control. 15 patients were enrolled, but one participant dropped-out after the first intervention - participants with available data: 14.
  SL: parallel design - SL sighted/SLblind/Sactivation/SLcontrol. OT: parallel design - OT real and OT control. MI: parallel design - MI real and MI control.
Measure: Mean (Standard Deviation); unit: microV
Arm/Group | Motor Learning (ML)-Sighted | Motor Learning -ML Blind | Motor Learning - ML Control | Somatosensory Learning (SL)- SL Sighted | Somatosensory Learning (SL)-SL Blind | Somatosensory Learning (SL)-SL Activation | Somatosensory Learning (SL)-SL Control | Observational Task (OT)- OT Real | Observational Task (OT)- OT Control | Mental Imagery (MI) - MI Real | Mental Imagery (MI) - MI Control
Number analyzed (Participants) | 14 | 14 | 14 | 10 | 10 | 10 | 10 | 15 | 15 | 14 | 15
microV
  Before | 1.37 (0.32) | 1.39 (0.25) | 1.28 (0.23) | 1.74 (0.78) | 1.67 (0.50) | 1.32 (0.29) | 1.30 (0.39) | 1.93 (0.75) | 1.79 (0.78) | 1.49 (0.81) | 1.70 (1.12)
  After | 1.27 (0.35) | 1.4 (0.28) | 1.49 (0.35) | 1.59 (0.73) | 1.47 (0.5) | 1.18 (0.39) | 1.28 (0.44) | 1.83 (0.74) | 1.65 (0.75) | 1.41 (0.81) | 1.66 (1.01)

ADVERSE EVENTS:
Arm/Group | Motor Learning (ML) Sighted | Motor Learning (ML) Blind | Motor Learning (ML) Control | Somatosensory Learning (SL) Sighted | Somatosensory Learning (SL) Blind | Somatosensory Activation (SA) | Somatosensory Learning (SL) Control | Observational Task (OT) - Real | Observational Task (OT) - Control | Mental Imagery (MI) - Real | Mental Imagery (MI) - Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/10 | 0/10 | 0/10 | 0/10 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/10 | 0/10 | 0/10 | 0/10 | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes